CLINICAL TRIAL: NCT03582514
Title: PreOperative Brain Irradiation in Glioblastoma
Acronym: POBIG
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: University of Liverpool (Other); The Netherlands Cancer Institute (Other); Northern Care Alliance NHS Foundation Trust (Other); University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFTSp200; 21/NW/0121 (Other: GM South Research Ethics Committee)
Record Dates: First submitted 2018-05-30; First posted 2018-07-11 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Glioblastoma Multiforme
Keywords: Radiotherapy; Preoperative; Neoadjuvant
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: The study uses a Continual Reassessment Method (CRM) to inform dose escalation and determine the MTD and MTIV. This is a Bayesian statistics-based model. It uses all available data from previous doses to guide dose escalation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose or volume radiation escalation (Experimental): Patients with a new radiological diagnosis of GBM (judged by the neuro-oncology multidisciplinary team) are to be considered for this study.
  This study arm will use 5 radiotherapy doses (6 Gy, 8 Gy, 10 Gy, 12 Gy and 14 Gy) and three treatment volumes (<30 cm3, 30-60 cm3 and >60 cm3). The study will use 6 dosing levels based on a combination of radiotherapy dose and treatment volume. The stepwise inclusion process allows for variation in tumour volume and location. The study will commence with dosing level 1: 8 Gy to <30 cm3 and 6 Gy to 30-60 cm3. In collaboration with the Clinical Trials Unit, the Trial Management Group will enter outcome data for patients at a given dose level into the CRM model. The model output will then guide dose escalation to determine the next dose level. After the single fraction of radiotherapy, patients will receive the standard treatment.
  Interventions: Radiation: Preoperative brain irradiation (single fraction)

INTERVENTIONS:
Radiation: Preoperative brain irradiation (single fraction) — Dose and volume escalation of preoperative single-fraction radiotherapy.

SUMMARY:
PreOperative Brain Irradiation in Glioblastoma (POBIG) is a phase I study that will test the safety and feasibility of a single fraction of preoperative radiotherapy in patients with a new radiological diagnosis of glioblastoma (GBM). After the single fraction of radiotherapy, patients will receive standard treatment. The standard treatment consists of resection of the tumor followed by (chemo)radiation (i.e. radiotherapy +/- daily temozolomide (75mg/m2) for 6 weeks (60Gy/30fr) or for 3 weeks (40Gy/15fr)).

DETAILED DESCRIPTION:
Glioblastoma is the most common primary malignant brain tumour in adults. Its outcomes are poor due to local disease progression in most patients. Current treatment includes surgery followed by chemotherapy and radiotherapy 4-6 weeks after surgery. In this time interval, some tumour cells do not receive any treatment. Furthermore, studies show that around half of all glioblastoma patients experience rapid early progression (REP) i.e. growth of the tumour in the time interval between surgery and postoperative chemotherapy/radiotherapy. REP is associated with a shorter survival and there are currently no effective treatments or preventative measures to address it. Radiotherapy delivered earlier before the operation could prevent REP and improve patient outcome. In this phase I study - PreOperative Brain Irradiation in Glioblastoma (POBIG), we will test the safety and feasibility of giving a single dose (fraction) of radiotherapy before surgery in patients with a new radiological diagnosis of glioblastoma. This study will be a dose escalation study to determine the maximum tolerated dose of preoperative radiotherapy and maximum volume of tumour that can be safely irradiated preoperatively. We hypothesise that preoperative radiotherapy will reduce the rate of REP and improve patient outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Male or female.
* New radiological diagnosis of glioblastoma.
* Performance status judged by World Health Organisation, Eastern Cooperative Oncology Group [ECOG] score = 0-1.
* Case has been reviewed by Neuro-oncology multidisciplinary team (MDT - neurosurgeon, clinical oncologist, radiologist and pathologist); MDT consensus that offering study entry is clinically appropriate and safe i.e. patient unlikely to come to harm (e.g. hydrocephalus) from delayed surgery and pre-operative radiotherapy based on available clinical information and imaging.
* Confirmation at first clinic visit that study entry is clinically appropriate and safe (e.g. lack of severe and debilitating symptoms of raised intracranial pressure).
* Intention to treat with surgical resection and postoperative adjuvant therapy as per current standard of care (Stupp regimen).
* Tumour size, location and configuration meet radiotherapy treatment planning criteria (e.g. to secure cold spot/hot spot, meets dose constraints for organs at risk when accounting for post-operative radiotherapy).
* Adequate haematological and biochemical parameters for surgery and contrast agent administration (full blood count and coagulation profile deemed acceptable by clinical team, eGFR >30ml/min).
* Mental capacity to consent for treatment.
* Able and willing to give informed consent.

Exclusion Criteria:

* Planned biopsy procedure only.
* Suspicion of other tumour on CT body scan or known malignancy except non-melanoma skin cancer, completely resected cervical or prostate cancer (with Prostate Specific Antigen of less than or equal to 0.1 ng/ml) within the past 3 years.
* Contraindications to contrast-enhanced MRI scanning (e.g. claustrophobia, gadolinium allergy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and maximum tolerated irradiation volume (MTIV) of single-fraction preoperative radiotherapy in patients with a new radiological diagnosis of glioblastoma | 18 months
  These will be determined by the following dose limiting complications:
  * Radiotherapy related swelling leading to a change of the scheduled date of surgery.
  * Post-operative radiotherapy commencement delayed to beyond 6 weeks after surgery due to radiation related symptoms and/or complications from surgery.
  * Interruption of post-operative radiotherapy >5 days.

SECONDARY OUTCOMES:
Registration of postoperative surgical complications. | 18 months
Radiotherapy related complications | 18 months
Progression free survival. | 18 months
Overall survival. | 18 months
Steroid dose after preoperative radiotherapy. | 18 months
The tumor volume differences measured between the post-surgery MRI and pre-radiotherapy MRI | 18 months
  To confirm usability of the MRI to select GBM patients for preoperative single fraction radiotherapy.
Concordance between MRI based diagnosis of glioblastoma and definitive histological diagnosis. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Gerben R Borst, MD, PhD, Principal Investigator — The Christie NHS Foundation Trust
Locations (1):
- The Christie NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

REFERENCES:
- [Derived] Waqar M, Roncaroli F, Djoukhadar I, Akkari L, O'Leary C, Hewitt L, Forte G, Jackson R, Hessen E, Withington L, Beasley W, Richardson J, Golby C, Whitehurst P, Colaco R, Bailey M, Karabatsou K, D'Urso PI, McBain C, Coope DJ, Borst GR. Study protocol: PreOperative Brain Irradiation in Glioblastoma (POBIG) - A phase I trial. Clin Transl Radiat Oncol. 2023 Jan 18;39:100585. doi: 10.1016/j.ctro.2023.100585. eCollection 2023 Mar. PMID 36845633